CLINICAL TRIAL: NCT06842043
Title: Clinical Effectiveness and Cost-Effectiveness of Real-Time Chest X-Ray Computer-Aided Detection System for Misplaced Endotracheal and Nasogastric Tubes and Pneumothorax in Emergency and Critical Care Settings
Brief Title: AI-Assisted Chest X-Ray for Misplaced Endotracheal and Nasogastric Tubes and Pneumothorax in Emergency and Critical Care Settings
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Fu Jen Catholic University Hospital (Other); Min-Sheng General Hospital (Other); National Taiwan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202412055DINA
Record Dates: First submitted 2025-02-12; First posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Endotracheal Tube; Nasogastric Tube; Pneumothorax
Keywords: Computer-aided detection system; Artificial intelligence; Pneumothorax diagnosis; Endotracheal tube; Nasogastric tube; Clinical effectiveness; Cost effectiveness
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Intervention Model Description: Each group requires 5,450 patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: AI-assisted model
- standard clinical practice (No Intervention)

INTERVENTIONS:
Other: AI-assisted model — physicians will be authorized to access the AI model's predictions during patient care as an additional decision-making reference. These predictions will be generated in seconds and can help identify issues such as tube misplacement (e.g., nasogastric tube, endotracheal tube) and pneumothorax through AI analysis of CXRs, which will alert the physician to review the images.
  Arms: Intervention

SUMMARY:
Background Advancements in artificial intelligence (AI) have driven significant breakthroughs in computer-aided detection (CAD) for chest X-ray imaging. National Taiwan University Hospital (NTUH) research team previously developed an AI-based emergency Capstone CXR system (MOST 111-2634-F-002-015-, Capstone project), which led to the creation of a chest X-ray module. This chest X-ray module has an established model supported by extensive research and is ready for direct application in clinical trials without requiring additional model training. This study will utilize three submodules of the system: detection of misplaced endotracheal tubes, detection of misplaced nasogastric tubes, and identification of pneumothorax.

Objective This study aims to apply a real-time chest X-ray CAD system in emergency and critical care settings to evaluate its clinical and economic benefits without requiring additional chest X-ray examinations or altering standard care and procedures. The study will evaluate the CAD system's impact on mortality reduction, post-intubation complications, hospital stay duration, workload, and interpretation time, alongside a cost-effectiveness comparison with standard care.

Methods This study adopts a pilot trial and cluster randomized controlled trial design, with random assignment conducted at the ward level. In the intervention group, units are granted access to AI diagnostic results, while the control group continues standard care practices. Consent will be obtained from attending physicians, residents, and advanced practice nurses in each participating ward. Once consent is secured, these healthcare providers in the intervention group will be authorized to use the CAD system. Intervention units will have access to AI-generated interpretations, whereas control units will maintain routine medical procedures without access to the AI diagnostic outputs.

Results The study was funded in September 2024. Data collection is expected to last from January 2025 to December 2027.

Conclusions This study anticipates that the real-time chest X-ray CAD system will automate the identification and detection of misplaced endotracheal and nasogastric tubes on chest X-rays, as well as assist clinicians in diagnosing pneumothorax. By reducing the workload of physicians, the system is expected to shorten the time required to detect tube misplacement and pneumothorax, decrease patient mortality and hospital stays, and ultimately lower healthcare costs.

ELIGIBILITY:
Inclusion Criteria for units:

* Emergency critical care or intensive care units.
* The units included the patients requiring chest X-rays due to endotracheal intubation, nasogastric tube insertion, or ventilator use with a risk of pneumothorax.

Exclusion Criteria for units:

* The unit supervisor doesn't agree to participate in the trial.
* The unit is unable to implement the AI-assisted system (e.g., no data connection or system support).

Inclusion Criteria for Patients:

● Patients who are adults and require chest X-ray due to one of the following conditions: endotracheal intubation, nasogastric intubation, or the use of a ventilator with the potential to cause pneumothorax.

Exclusion Criteria for Patients: Patients in isolation wards or pediatric

* Patients in isolation wards.
* Patients in Infant Intensive Care Unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10900 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
In-hospital Mortality | During the hospital stay, an average of 1 week
  The patient's survival is monitored after undergoing a chest X-ray until hospital discharge.

SECONDARY OUTCOMES:
Length of Hospital Stay | During the hospital stay, an average of 1 week
  The time a patient spends in the hospital from admission to discharge, usually measured in days.
Misplacement Detection Time | During the hospital stay, an average of 1 week
  Evaluates whether the AI system can reduce the time to detect misplaced catheters or pneumothorax, thereby improving the timeliness of clinical intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan